CLINICAL TRIAL: NCT04090905
Title: Incidence of Post-operative Atrial Fibrillation Secondary to Abdominal Surgery - A Single-centre, Prospective, Cohort Study
Brief Title: Incidence of Post-operative Atrial Fibrillation Secondary to Abdominal Surgery
Acronym: SECAFIB-SURG
Status: Completed | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Christoffer Valdorff Madsen, Primary Investigator, Frederiksberg University Hospital
Other Study IDs: H-19033464
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation; Surgery--Complications
Keywords: post-operative atrial fibrillation; abdominal surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unselected cohort: Consecutive adult patients who were referred for acute abdominal surgery. Patients underwent standard observation in either a surgical ward (utilizing the National Early Warning Score) or the intensive care unit with continuous respiratory and circulatory monitoring.
  Interventions: Other: Standard clinical monitoring
- Subgroup with Holter monitoring: Consecutive adult patients who were referred for acute abdominal surgery in the time interval 7 AM to 11 PM. Holter monitoring was applied on top of standard observation in either a surgical ward (utilizing the National Early Warning Score) or the intensive care unit with continuous respiratory and circulatory monitoring.
  Interventions: Other: Standard clinical monitoring; Diagnostic Test: Holter monitoring

INTERVENTIONS:
Other: Standard clinical monitoring — Standard observation in either a surgical ward (utilizing the National Early Warning Score) or the intensive care unit with continuous respiratory and circulatory monitoring.
Diagnostic Test: Holter monitoring — Cardiac rhythm monitoring before, during, and until hospital discharge (preferably ≥72 hours after abdominal surgery)
  Groups: Subgroup with Holter monitoring

SUMMARY:
Background and purpose Post-operative AF (POAF) is considered a phenomenon rather than a definite diagnosis and the current clinical guidelines have no specific recommendations regarding its management. Few prospective studies have been performed in non-cardiac conditions and the consequences of POAF in patients without known heart disease are not well described. However, recent data suggest an association between POAF in relation to non-cardiac surgery and increased post-operative mortality and stroke. POAF in relation to abdominal surgery seems common (incidence: 8-18%); however, the true incidence is uncertain. The available studies are few, heterogeneous, and often methodologically inadequate. The study aims at reporting the incidence of atrial fibrillation (AF), and associated complications, in relation to abdominal surgery.

Material and methods Designed as a prospective, single-centre, cohort study of consecutive adult patients undergoing acute* abdominal surgery at the Department of Abdominal Surgery at Bispebjerg Hospital. Patients who are pregnant or where follow-up is not possible will be excluded. Patients will be examined pre-operatively by ECG and signal processed surface ECG (wavECG). A subset of patients admitted to the Department in the time interval of 7 AM to 11 PM$, will be offered heart rhythm monitoring from admission and until discharge (preferably ≥72 hours post-operatively). Additional follow-up will be based on a review of patient charts at discharge and one# month postoperatively. The primary endpoint is the occurrence/recurrence of AF. The study will include 400-500 patients of which an estimated 2/3 will wear heart rhythm monitoring corresponding to 264-330 patients.

Perspective If more thorough heart rhythm monitoring of patients undergoing abdominal surgery leads to the identification of more patients with AF, routine continuous heart rhythm monitoring should be considered recommended in upcoming guidelines to prevent associated complications.

Footnote(s): See 'Detailed Description' below.

DETAILED DESCRIPTION:
Background and rationale Post-operative AF (POAF), i.e. atrial fibrillation (AF) that occurs secondarily to surgery is considered a phenomenon rather than a definite diagnosis, and continuous anti-coagulation is not recommended in AF of short duration and non-persistent AF.1,2 The most recent guidelines from the European and American Societies of Cardiology have no specific recommendation regarding the management of secondary AF, though referral to an outpatient cardiology clinic can be considered if the condition is not self-limiting.3,4 Despite this, recent data from the Framingham population suggest that secondary AF is not a benign condition,5,6 and some studies have found POAF in relation to non-cardiac surgery to be associated with increased post-operative mortality and stroke.7-9 Currently few prospective studies have been performed in non-cardiac conditions and the consequences of secondary AF in patients without known heart disease are not well described. POAF in relation to non-cardiac surgery is common with an average incidence of 10.94%.10 However, the true incidence of POAF in relation to non-cardiac surgery is uncertain, as the available studies are few, heterogeneous, and often methodologically inadequate.10 Different risk-stratification models exist, however it is still challenging to accurately predict which patients will develop AF both perioperatively and in the years following surgery.11-14 Important risk factors for developing POAF are: age (age 65-74, OR 2.08; age >85, OR 3.56), hypertension (OR 3.66), heart failure (OR 1.64), thyroid disease (OR 6.29), laparotomy vs laparoscopy (OR 3.30) and duration of surgery (> 600 min, OR 1.38).10 The use of electrocardiogram (ECG) in risk stratification for AF and stroke is not yet incorporated in clinical guidelines. However, short and prolonged p-wave and p-wave terminal force in lead V1 (PTFV1) is correlated with AF.15 Myovista (HeartSciences, Southlake, Texas, USA) is a novel ECG utilizing continuous wavelet transform signal processing (wavECG) and can be used to prove left ventricular diastolic dysfunction (LVDD).16 LVDD is in other studies associated with AF.17-20 These new biomarkers might improve the identification of patients at risk of developing POAF.

Purpose The study aims at reporting the incidence of AF, and associated complications, in relation to acute abdominal surgery. Concurrently, patients will be characterized by specialized ECG analysis and wavECG.

Methods Prospective, single-centre, cohort study of consecutive patients undergoing acute* abdominal surgery. Patients will be identified among acute referrals for the Department of Abdominal Surgery at Bispebjerg-Frederiksberg Hospital. The Investigator (Department of Cardiology at Bispebjerg-Frederiksberg Hospital) will ensure signed informed consent prior to any study-related examinations. Surgery will be performed at the Department of Abdominal Surgery at Bispebjerg-Frederiksberg Hospital independently of study enrolment. A subset of patients will be enrolled in a feasibility study of continuous cardiac rhythm monitoring (C3+, Cortrium, Copenhagen, Denmark). Heart rhythm monitoring will be worn from admission and until discharge (preferably ≥72 hours post-operatively) in patients admitted to the Department in the time interval of 7 AM to 11 PM$. Additional follow-up will be based on a review of patient charts at discharge and one# month postoperatively.

No randomization or placebo will be used. ECG measurements will be compared to existing data from a healthy population.

Measurements

* ECG: AF, PR-interval, p-wave area, PTFV1
* wavECG: LVDD
* Heart rhythm monitoring: AF

Statistical considerations Consecutive patients attending the Department of Abdominal Surgery at Bispebjerg-Frederiksberg Hospital will be invited to participate in the pre- and post-operative examination programme. The study's aim is to identify the incidence of peri- and postoperative AF. Hence, sample size calculations are uncertain. The expected incidence of AF for patients undergoing non-oesophageal abdominal surgery is at least 7.63%.10 Pre-operative p-wave indices have shown the ability to predict POAF in a cardiac surgery population of 105 patients (with a POAF incidence of 11%).21 wavECG has been used to show LVDD in a study population of 188 patients referred for computed tomography angiography of the heart.16 The study will include 400-500 patients of which an estimated 2/3 will wear heart rhythm monitoring corresponding to 264-330 patients. Follow-up will be one month.

Normality was inspected visually by histograms and tested by Shapiro-Wilk. Nonparametric statistics were used. Wilcoxon rank-sum (continuous variables) and Chi-square and Fisher's exact test (categorical variables) were used as appropriate. Data were presented as median with interquartile range (IQR) for continuous variables and frequency with percentages for categorical variables. Odds ratios (OR) with 95% confidence intervals (CI) were calculated for dichotomous values by univariate logistic regression. Multiple logistic regression was used to adjust for variables' influence on the primary outcome of POAF and the secondary outcome of severe adverse events. Based on an á priori knowledge of risk factors of atrial fibrillation and expected important surgical factors, variables were chosen for the full multivariate model. The following variables were included: age, sex, prior atrial fibrillation, prior stroke, hypertension, heart failure, heart valve disease, chronic renal disease, diabetes mellitus, vascular disease, chronic obstructive pulmonary disease, cancer, surgery invasiveness, and surgery urgency. For multivariate modeling of the secondary outcome, POAF was added to the full model as it was expected to influence the development of the outcome. Subsequently, the full multivariate logistic regression model was reduced to a prediction model. Variables with p<0.05 remained in the prediction model, while variables with p>0.05 were eliminated. Multicollinearity was checked and a Variance Inflation Factor level <5 was accepted. McFadden's R-squared test was applied to evaluate model fit, while Analysis of variance (ANOVA) tests were applied to compare the components of the model, to reduce the risk of overfitting. A receiver operating characteristic curve (ROC) with area under the curve (AUC) was calculated for the multivariate model. The Closest Topleft decision rule was applied to define the optimal sensitivity and specificity values. For AUC, sensitivity, and specificity, 95% confidence intervals were produced through bootstrapping with 2000 replicates. All tests were two-sided, and a p< 0.05 was considered statistically significant. RStudio (version 1.4.1717) was used for statistical analyses.

Footnote(s): *The study was originally designed to include both acute and elective patients, but due to limited availability of heart rhythm monitoring devices, prior to study initiation (June 5, 2020), we decided to enroll patients referred for acute abdominal surgery only. $The study was originally planned to apply heart rhythm monitors all 24 hours of the day. This was not possible due to logistics, and prior to study initiation, we agreed to apply monitoring to all patients admitted between 7 AM to 11 PM. #The study was originally planned for 12 months follow-up but was reduced to one month, due to limitations of the permissions achieved prior to study initiation. In addition, an outpatient clinic visit 3 months after surgery was planned where ECG and heart rhythm monitor examinations were to be repeated. The visits were canceled due to local COVID-19 restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Acute abdominal surgery (non-oesophageal)
* Age ≥ 16 years

Exclusion Criteria:

* Pregnancy
* Follow-up not possible

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult patients undergoing acute abdominal surgery at the Department of Abdominal Surgery at Bispebjerg Hospital (Copenhagen, Denmark)
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of clinically recognized peri- and post-operative atrial fibrillation | In-hospital, defined as occurring from termination of surgery and until discharge from the hospital. Assessed up to 7 days from surgery.
  Occurrence of clinically recognized POAF, defined as recognized by clinical staff and verified by a 12-lead electrocardiogram and adjudicated by Cardiology specialists.

SECONDARY OUTCOMES:
Incidence of peri- and post-operative atrial fibrillation by cardiac rhythm monitoring | In-hospital, defined as occurring from termination of surgery and until discharge from the hospital. Assessed up to 7 days from surgery.
  Atrial fibrillation (AF) lasting more than 30 seconds on cardiac rhythm monitoring was sufficient for an AF diagnosis.
Incidence of clinically recognized post-operative atrial fibrillation | Out-of-hospital, defined as within 30 days from index surgery
  Occurrence of clinically recognized POAF, defined as recognized by clinical staff and verified by a 12-lead electrocardiogram and adjudicated by Cardiology specialists.
Incidence of clinical events after surgery | In-hospital, defined as occurring from termination of surgery and until discharge from the hospital. Assessed up to 7 days from surgery.
  Clinical events defined as: death, life-threatening complications, major abdominal reoperation, prolonged hospitalization (admissions with complications requiring hospitalization beyond standard treatment)
Incidence of clinical events after surgery | Out-of-hospital, defined as within 30 days from index surgery
  Clinical events defined as: death, life-threatening complications, major abdominal reoperation, prolonged hospitalization (admissions with complications requiring hospitalization beyond standard treatment), or hospital readmission.
Number of patients with abnormal p-wave indexes | Before surgery
  Abnormal p-wave indexes on electrocardiogram
Number of patients with left ventricular diastolic dysfunction | Before surgery
  Left ventricular diastolic dysfunction as measured on wavECG (Myovista)

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer V Madsen, MD, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided